CLINICAL TRIAL: NCT04609605
Title: Assessment of Right Ventricular Function After Acute Pulmonary Embolism Using Speckle Tracking Echocardiography
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Said Rashwan, doctor, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: speckle tracking in PE
Record Dates: First submitted 2020-10-26; First posted 2020-10-30 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with acute pulmonary embolism (Experimental): speckle tracking echocardiography for patient with acute pulmonary embolism
  Interventions: Device: speckle tracking echocardiography

INTERVENTIONS:
Device: speckle tracking echocardiography — speckle tracking echocardiography of right ventricle

SUMMARY:
1. To asses regional RV function in patients presented with acute pulmonary embolism using speckle tracking echocardiography
2. To evaluate its relationship to long term mortality.

DETAILED DESCRIPTION:
Pulmonary embolism (PE) is the third most common cardiovascular cause of death after myocardial infarction and stroke . The incidence of PE has been increasing ,with significant associated mortality; a recent registry of PE patients reported a mortality rate > 10% at 30 days. There are a number of emerging contemporary PE therapies, including thrombolysis, catheter intervention and surgery. Early and accurate identification of PE in patients is therefore critical. A transthoracic echocardiogram (TTE) may help when there is a clinical suspicion for PE, and its use in confirmed PE is widely recommended . A number of right atrial (RA) and right ventricular (RV) parameters have been shown to be abnormal in patients with PE . In addition, RA and RV enlargement portends a worse prognosis in these patients .

ELIGIBILITY:
Inclusion Criteria:

1. clinical diagnosis of acute pulmonary embolism
2. Age: 20 - 70 years.

Exclusion Criteria:

1. coronary artery disease
2. patient of Atrial fibrillation.
3. Patient of impaired RV function due to chest disease (Cor-pulmonale)
4. patient with impaired Ejection fraction (EF) <50%
5. Moderate to severe valvular heart disease.
6. Atrio-ventricular conduction disturbance.
7. Poor echogenicity

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
improve management of acute pulmonary embolism | baseline
  comparison between speckle tracking echocardiograpgy and conventional echocardiography in pulmonary embolism

REFERENCES:
- [Background] Wendelboe AM, Raskob GE. Global Burden of Thrombosis: Epidemiologic Aspects. Circ Res. 2016 Apr 29;118(9):1340-7. doi: 10.1161/CIRCRESAHA.115.306841. PMID 27126645
- [Background] McConnell MV, Solomon SD, Rayan ME, Come PC, Goldhaber SZ, Lee RT. Regional right ventricular dysfunction detected by echocardiography in acute pulmonary embolism. Am J Cardiol. 1996 Aug 15;78(4):469-73. doi: 10.1016/s0002-9149(96)00339-6. PMID 8752195
- [Background] Fields JM, Davis J, Girson L, Au A, Potts J, Morgan CJ, Vetter I, Riesenberg LA. Transthoracic Echocardiography for Diagnosing Pulmonary Embolism: A Systematic Review and Meta-Analysis. J Am Soc Echocardiogr. 2017 Jul;30(7):714-723.e4. doi: 10.1016/j.echo.2017.03.004. Epub 2017 May 9. PMID 28495379
- [Background] Trivedi SJ, Altman M, Stanton T, Thomas L. Echocardiographic Strain in Clinical Practice. Heart Lung Circ. 2019 Sep;28(9):1320-1330. doi: 10.1016/j.hlc.2019.03.012. Epub 2019 Apr 12. PMID 31064715